CLINICAL TRIAL: NCT01813370
Title: A Registry for Patients Treated on the Clinical Trial TAX 3503 (A Randomized, Open Label, Multicenter, Phase III, 2-Arm Study of Androgen Deprivation With Leuprolide, +/- Docetaxel for Clinically Asymptomatic Prostate Cancer Subjects With a Rising PSA Following Definitive Local Therapy)
Brief Title: A Registry for Patients Treated on the Clinical Trial TAX 3503
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Laval University (Other); Vancouver General Hospital (Other); London Health Sciences Centre (Other); Centre Hospitalier Universitaire de Montreal - Hospital Notre-Dame (Unknown); Princess Margaret Hospital, Canada (Other); CancerCare Manitoba (Other); Tom Baker Cancer Centre (Other); Urocentrum Praha s.r.o. (Unknown); Fakultní nemocnice Na Bulovce (Unknown); Hospital Jablonec nad Nisou, p.o (Unknown); Klaipėda University (Other); Lithuanian University of Health Sciences (Other); Oncology Institute of Vilnius University (Unknown); Fakultna Nemocnica s poliklinikou J.A. Reimana Presov, Klinika urologie (Unknown); Martinska Fakultna Nemocnica, Urologicke klinika (Unknown); Fakultna nemocnica s poliklinikou (Unknown); BratislavaNemocnica ak. L Derera, Urologicka klinika (Unknown); Urologic Consultants of Southeastern PA (Other); Columbia University (Other); GU Research Network, LLC (Other); Carolina Urologic Research Center (Other); Lancaster Urology (Unknown); Kansas City Veteran Affairs Medical Center (U.S. Federal Agency); Urology San Antonio Research PA (Unknown); University of Texas Southwestern Medical Center (Other); University of Cincinnati (Other); St. Alexius Medical Center Clinical Research Services (Unknown); Barbara Ann Karmanos Cancer Institute (Other); Johns Hopkins University (Other); Duke University (Other); Vanguard Urologic Research Foundation (Other); The Urological Institute of Northeastern NY (Unknown); Urology Associates Medical Group (Unknown); Hospital de Sabadell (Other); Lahey Clinic (Other); San Bernardino Urological Associates (Unknown); Columbus Urology (Unknown); Niepubliczny Specjalistyczny Onkologiczny Zaklad Opienki Zdrowotnej (Unknown); Vinzenzkrankenhaus Hannover, Urologische Abteilung (Uro-Onkologie) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 12-225
Record Dates: First submitted 2013-03-13; First posted 2013-03-19 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Prostate Cancer
Keywords: TAX 3503; MSKCC IRB#07-101; 12-225
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples With DNA — Serum PSA evaluations Serum testosterone levels

GROUPS / COHORTS (1):
- Pts with prostate cancer: Patients who have progressed or hit their 36 month post treatment date between the closure of TAX3503 and the activation of this TAX3503 Registry protocol will be permitted on the study to capture their date of progression or their 36 month post treatment progression free date.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention is planned as part of this protocol. Historical data will be transferred to MSK via electronic data transfer. Patient's PSA, testosterone, and vital status data will be transferred to MSK via electronic data transfer.

SUMMARY:
The purpose of this study is to continue follow-up on patients who were treated on the study called TAX 3505 (MSK IRB #07-101). The sponsor of this study, has decided to end the study early, before all patients have completed all planned follow-up tests. As a result, the investigators do not yet know whether hormonal therapy alone, or in combination with docetaxel, is better at preventing prostate cancer recurrence in patients who had a rising PSA after prostatectomy. This study will continue following patients according to a schedule that is similar to that found in the TAX 3503 (MSK IRB #07-101) study in order to answer that question. This study is known as a registry study. The patients' will not receive any treatment as part of this study. Instead, they will be asked to have a blood test performed once every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The registry will include the database of all patients registered to TAX3503. Those patients who will be prospectively tracked through the registry are those who meet the following criteria:

  1. The patient must have been registered to TAX3503
  2. The patient must not have met the definition of progression as defined in TAX3503 while on TAX3503 Patients who have progressed or hit their 36 month post treatment date between the closure of TAX3503 and the activation of this TAX3503 Registry protocol will be permitted on the study to capture their date of progression or their 36 month post treatment progression free date.

Exclusion Criteria:

* Patients who were not registered to TAX3503 are not eligible to have their data stored in this registry.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are presently on TAX3503 and undergoing followup for evidence of progressive disease will be approached by their study physicians at their local sites to enter the registry. No other patient will be approached or recruited. Some sites that were part of the TAX3503 study are unable to open this registry at their site. In order to minimize the number of participants whose information might be lost, Memorial Sloan-Kettering Cancer Center (MSKCC) will inform these sites that they may refer their participants to MSKCC for this registry.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2013-03; Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
progression free survival | 1 year
  For patients treated on TAX3503 that will enable the study to achieve its primary endpoint of comparing the efficacy of its treatment arms as determined by progression-free survival during the period from randomization to progression or death or last followup.

SECONDARY OUTCOMES:
annotating clinical outcomes | 1 year
  To utilize this registry for the purposes of annotating clinical outcomes to the biospecimens collected under TAX3503.
overall survival differences | 1 year
  Between the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Michael Morris, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (5):
  - John Hopkins Medical Center, Baltimore, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Urological Associates of Lancaster, Lancaster, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
- Cancer Care Manitoba, Winnipeg, Manitoba, Canada
- Lithuania (2):
  - Hospital of Lithuanian University Health Sciences Kauno Klinikos, Kaunas, Klinikos
  - Klaipeda University Hospital, Klaipėda

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/